CLINICAL TRIAL: NCT04851795
Title: Effectiveness of a Supervised Hospital-based Physical Exercise Intervention to Reduce Stress in Health Care Professionals
Brief Title: Effectiveness of a Supervised Hospital-based Physical Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bioaraba Health Research Institute (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PA01
Record Dates: First submitted 2021-04-15; First posted 2021-04-20 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Stress, Psychological; Anxiety
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supervised physical exercise sessions (Experimental): Participants assigned to the supervised exercise group will perform a supervised routine of approximately 30 minutes, 2 days per week (Monday and Wednesday at the Txagorritxu hospital, and Tuesday and Thursday at the Santiago hospital from 7:15 to 7:45 and from 15:15 to 15:45).
  Interventions: Other: supervised physical exercise sessions
- unsupervised physical exercise sessions (Other): For the non-supervised group, we will propose climbing the stairs from floor 0 to floor 7 three times during the working day and doing planks and stretching exercises outside of work. For the latter, an educational session will be given at the beginning of the study to explain how to perform them correctly.
  Interventions: Other: unsupervised physical exercise

INTERVENTIONS:
Other: supervised physical exercise sessions — Participants assigned to the supervised exercise group will perform a supervised routine of approximately 30 minutes, 2 days per week (Monday and Wednesday at the Txagorritxu hospital, and Tuesday and Thursday at the Santiago hospital from 7:15 to 7:45 and from 15:15 to 15:45).
  Arms: supervised physical exercise sessions
Other: unsupervised physical exercise — For the non-supervised group, we will propose climbing the stairs from floor 0 to floor 7 three times during the working day and doing planks and stretching exercises outside of work. For the latter, an educational session will be given at the beginning of the study to explain how to perform them correctly.
  Arms: unsupervised physical exercise sessions

SUMMARY:
To assess if physical activity is effective in reducing stress and anxiety in healthcare professionals.

DETAILED DESCRIPTION:
To assess if physical activity is effective in reducing stress and anxiety in healthcare professionals.

To evaluate if physical activity is effective in improving the physical and mental state of health care professionals and improving several blood parameters (lipid profile and blood glucose).

ELIGIBILITY:
Inclusion criteria

* Apt for sports practice after review by the corresponding health professional of the Occupational Health Service,
* Motivation for sports practice (could be self-referred or on an EVA scale from a score for example of 6) being 0 not motivated at all and 10 totally motivated.

One could extrapolate the score limits of the EVA scale pain no motivation=0; mild motivation=1,2; moderate=3-5; high from 6.

* Professionals whose working day does not coincide with the hours during which the sessions are to be given.
* Professionals who do not work shifts.

Exclusion Criteria:

* Any type of contraindication for sports practice (Annex I),
* Staff who, due to their activity, have greater mobility in the hospital (orderlies).
* Osteoarticular injuries, cervical and lumbalgias.

Withdrawal criteria

-Within the intervention group - absence maximum two weeks to the exercises. This will not be taken into account during the summer period.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress | at six months
  Perceived stress scale-PSS. PSS scores are obtained by inverting the responses (e.g. 0 = 4, 1 = 3, 2 = 2, 3 = 1 and 4 = 0) to the four positive items (items 4, 5, 7 and 8) and then adding up all the points on the scale.

SECONDARY OUTCOMES:
Goldberg anxiety questionnaire | at six months
  Goldberg anxiety questionnaire. This questionnaire has a total of 9 items. A score greater than or equal to 4 is indicative of anxiety.
Short Form Survey_Mental health | at six months
  Mental component of the SF12 questionnaire. For each of the 8 dimensions, the items are coded, aggregated and transformed into a scale ranging from 0 (worst health status for that dimension) to 100 (best health status). The number of response options ranges from three to six, depending on the item.
Short Form Survey_Physical condition | at six months
  Physical component of the SF12 questionnaire. For each of the 8 dimensions, the items are coded, aggregated and transformed into a scale ranging from 0 (worst health status for that dimension) to 100 (best health status). The number of response options ranges from three to six, depending on the item.
Ruffier index | at six months
  The Ruffier test is a test performed to measure short-term aerobic endurance and cardiac recovery capacity, and therefore the level of physical fitness in individuals. An index below 0 indicates a good physical condition. Its average value is between 5 and 10. Above 10 the patient is considered to have a poor adaptation to exertion.
Weight | at six months
  Weight
Body mass index | at six months
  Body mass index
lipid profile | at six months
  Colesterol, HDL, LDL, triglycerides
glycosylated hemoglobin | at six months
  glycosylated hemoglobin
work absenteeism | at six months
  work absenteeism

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Araba university hospital, Vitoria-Gasteiz, Alava
  - Bioaraba Health Research Institute, Vitoria-Gasteiz, Alava

IPD SHARING:
Plan to Share IPD: No